CLINICAL TRIAL: NCT04889989
Title: A Single-Arm, Prospective, Multicenter Study to Evaluate the Effectiveness and Safety of the NeuWave Certus Microwave Ablation System in Chinese Patients With Primary or Secondary Tumors in the Lung
Brief Title: Microwave Ablation in Chinese Patients With Lung Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in company strategy.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU_2020_02
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cancer of the Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective, multicenter clinical trial with a performance goal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microwave Ablation of Lung Tumor (Other): Adult patients with non-small cell lung cancer (NSCLC) or oligometastatic lung tumors who plan to receive percutaneous microwave ablation.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Microwave Ablation — Percutaneous microwave ablation using the NeuWave Microwave Ablation System for non-small cell lung cancer or oligometastatic lung tumors

SUMMARY:
Adult patients with non-small cell lung cancer (NSCLC) or oligometastatic lung tumors will all receive microwave ablation (MWA) performed percutaneously by doctors who are experienced in lung tumor ablation. 120 patients will participate across 8 clinical study sites all in China.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form and willing to fulfill the study-related assessments and procedure schedule.
2. Lung tumor patients ≥ 18 years of age who are ineligible for/decline surgery and who plan to receive microwave ablation therapy.
3. ECOG performance status score of 0-2.
4. Patients with stages IA1-IA2 NSCLC with documented results from a biopsy or patients with clinically diagnosed oligometastatic lung tumor.
5. Tumor(s) to be ablated in a single surgery should be a maximum of one NSCLC tumor or a maximum of three ipsilateral oligometastatic lung tumors.
6. Tumor(s) to be ablated in a single surgery should be ≤ 2cm, locate in the outer two-thirds of a lung, not closer than 1 cm from the hilum of lung, great vessels, principal bronchus, trachea or esophagus, and not contiguous with the pleura.

Exclusion Criteria:

1. Pregnant or breast-feeding.
2. Patients with implantable pacemakers or other electronic implants.
3. Oligometastatic tumors patients whose primary lesion cannot be controlled or have widely metastases, in the opinion of the investigator and/or treating oncologist.
4. Any planned concurrent procedure at the time of ablation.
5. Planned treatment for other tumors in the same side lung during the study period.
6. With a skin infection or ulceration at the site to be punctured by probe(s).
7. Clinical or imaging findings consistent with an active pulmonary infection.
8. Patients with severe pulmonary fibrosis in the area intended to ablate, especially drug-induced pulmonary fibrosis.
9. Patients with prior radiotherapy in the area intended to ablate.
10. Patients with uncontrolled malignant pleural effusion at the lung side with tumor to ablate.
11. Tumors where the anticipated zone of ablation would encompass significant (in the opinion of the treating physician) emphysematous or bullous disease.
12. The investigator anticipates that the ablation zone of the multiple tumor(s) to be ablated may have overlapping ablation zones.
13. Patients who have received lung ablation or surgical resection therapy within 30 days prior to the ablation procedure under study and those who plan to receive lung tumor ablation or surgical resection therapy or radiation therapy on the ablated lung side before completing the primary efficacy endpoint assessment approximately 30 days after the ablation procedure.
14. Patients who received systemic therapy such as chemotherapy, targeted drug therapy, or immunotherapy within 7 days prior to the ablation procedure under study, and patients who had a systemic treatment plan such as chemotherapy, targeted drug therapy, immunotherapy, etc. before completing the primary efficacy endpoint assessment approximately 30 days after the ablation procedure.
15. Patients with uncorrectable coagulopathy based on investigator judgment.
16. Patients with a platelet count ≤ 50 × 109/L.
17. Patients who cannot discontinue antiplatelet medication (e.g., aspirin, clopidogrel, prasugrel, ticagrelor) at least 5 days before the ablation procedure through 24 hours post-procedure.
18. Patients who cannot discontinue anticoagulant medication (e.g., rivaroxaban, apixaban, dabigatran, edoxaban) at least 3 days before the ablation procedure through 24 hours post-procedure.
19. Patients who cannot discontinue warfarin before at least 5 days before the ablation procedure of the study or have an INR > 1.5.
20. As judged by the investigator, the patient has hypertension that cannot be effectively controlled by pharmacological treatments.
21. Severe hepatic, renal, cardiac, pulmonary or cerebral insufficiency, severe anemia, dehydration, and severe nutrition and metabolism disorders, which cannot be corrected or improved within a short term; or serious systemic infection; or severe neuromuscular diseases.
22. Expected survival less than 6 months.
23. Participation in any other interventional clinical study within 30 days before screening.
24. Physical or psychological condition which would impair study participation.
25. Patient is judged unsuitable for study participation by the investigator for any other reason.

    Intra-Ablation Exclusion Criteria:
26. Before ablation probe puncture on the skin, patient is judged unsuitable for study participation due to intolerance to anesthesia.
27. Before ablation probe puncture on the skin, patient is judged unsuitable for study participation due to presenting any other condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Hospital, Beijing
  - Pecking University Shenzhen Hospital, Beijing
  - The First Affiliated Hospital of Fujian Medical University, Fujian
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Henan Cancer Hospital, Henan
  - Hunan Cancer Hospital, Hunan
  - Qilu Hospital of Shandong University, Shandong
  - Fudan University Shanghai Cancer Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chinese adult patients with NSCLC (non-small cell lung cancer) or oligometastatic lung tumors (2cm or less in size) who were candidates for percutaneous microwave ablation were considered for the study. Patients were given the Informed Consent Form to read, ask questions, and sign prior to any study procedures being performed or data being collected.
Pre-assignment Details: As a single-arm study, all patients enrolled received the same treatment: microwave ablation using the NEUWAVE Microwave Ablation System and Probes.
  The first 2 patients at each treating site (2 patients at 2 sites = 4 total patients) were part of the 'run-in' cohort. The Run-In cohort was implemented to reduce operational bias due to the learning curve. Run-In patients were included in the safety analysis set only.
Units Other Than Participants: Tumors
Groups:
- Microwave Ablation: Lung tumors treated with microwave ablation (includes the run-in patients) and still alive at the end of the study (1-year post-ablation)
Period: Overall Study
Arm/Group | Microwave Ablation
Started (13) | 13; 14 Tumors (Same as the number of patients/tumors treated and is the number used for all safety analyses (like AE/SAE reporting).)
Run-In (4) | 4; 4 Tumors (Run-in patients only included in the safety analysis.)
Withdrew Consent (Withdrew consent after being treated and before the 1-month follow-up visit.) | 1; 1 Tumors
Died | 1; 1 Tumors
Lost to Follow-Up | 1; 2 Tumors
Completed (6) | 6; 6 Tumors
Not Completed | 7; 8 Tumors

BASELINE CHARACTERISTICS:
Population: The 9 baseline participants is calculated from the 13 patients who were treated with microwave ablation minus the 4 run-in patients (13-4=9).
  The 9 baseline patients had 10 tumors treated.
Units Other Than Participants: Tumors
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 9
Number analyzed (Tumors) | 10
Age, Continuous [Median (Full Range); unit: Years] | 54.0 [44 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Technical Efficacy Rate
Description: Percentage of tumors that were completely covered by the ablation zone with no sign of pathological enhancement according to the lung contrast-enhanced CT assessment as assessed by the Independent Review Committee.
Time Frame: 30 days (+/- 7 days) post-ablation
Measure: Count of Units; unit: Tumors
Units Other Than Participants: Tumors
Groups:
- Microwave Ablation: Lung tumors treated with microwave ablation (does not include the run-in patients)
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 8
Number analyzed (Tumors) | 9
Tumors | 8

2. Secondary Outcome: Technical Success Rate
Description: Percentage of tumors that achieve A0 or A1 ablation classification determinations (i.e., complete tumor ablation with a surrounding margin) based on the lung CT immediately following the initial ablation procedure and as assessed by the Independent Review Committee.
Time Frame: Ablation Day (day 0)
Measure: Count of Units; unit: Tumors
Units Other Than Participants: Tumors
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 8
Number analyzed (Tumors) | 9
Tumors | 9

3. Secondary Outcome: Local Tumor Progression
Description: Progression of disease to a tumor treated during the original microwave ablation procedure.
Time Frame: 1 year post-ablation
Measure: Count of Units; unit: Tumors
Units Other Than Participants: Tumors
Groups:
- Microwave Ablation: Lung tumors treated with microwave ablation (does not include the run-in patients) with 1-year follow-up.
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 7
Number analyzed (Tumors) | 8
Tumors | 1

4. Secondary Outcome: Overall Survival
Description: Rate of patients still alive 1-year post-ablation (includes lead-in participants so out of 13).
Time Frame: 1-year post-ablation
Measure: Count of Participants; unit: Participants
Groups:
- Microwave Ablation: Lung tumors treated with microwave ablation (includes the run-in patients)
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 13
Participants | 12

5. Secondary Outcome: Progression-Free Survival
Description: Rate of patients still alive 1-year post-ablation without any sort of progression of disease (local, regional, or distant).
Time Frame: 1-year post-ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 12
Participants | 10

ADVERSE EVENTS:
Time Frame: 1-year post-ablation
Description: From the time of the ablation procedure through 30 days post-ablation, all AEs and serious AEs (SAEs) were recorded. After 30 days post-ablation, only AEs judged by the PI as related to the study device and/or procedure and all SAEs were reported.
  AEs/SAEs summarized below include all events reported and do not distinguish between being device- or procedure-related.
Groups:
- All Patients Treated With Microwave Ablation: Includes all patients treated with microwave ablation (including run-in patients)
Arm/Group | All Patients Treated With Microwave Ablation
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Treated With Microwave Ablation (N=13)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Treated With Microwave Ablation (N=13)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
The study was originally statistically powered and planned to enroll/treat 120 patients. However, the study was terminated early after a change in Sponsor strategy. Only 13 patients (4 being run-in) across 2 sites were enrolled and treated. All results provided are descriptive in nature only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have the first right to publish the study data. If publication of the study data by the Sponsor has not occurred within eighteen (18) months of study completion/termination, the PI may publish the results from the PI his/her site individually. The PI should provide the Sponsor with at least thirty (30) days for review of the publication.

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04889989/Prot_002.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04889989/SAP_003.pdf